CLINICAL TRIAL: NCT02460523
Title: Management and Outcome of Borderline Common Bile Duct With Stone
Brief Title: Management of Borderline Common Bile Duct Stone
Acronym: CBDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, Gastroenterology surgical center, mansoura university, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: borderline CBDS
Record Dates: First submitted 2015-05-22; First posted 2015-06-02 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2012-04

CONDITIONS: Common Bile Duct Stone
MeSH Terms: conditions — Gallstones | interventions — Conservative Treatment; Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- conservative (Active Comparator): 1- Patients in conservative treatment group will receive medical treatment in the form of antibiotics (3rd generation cephalosporine), analgesics (NSAID eg Ibuprofen ) and antispasmodics for 3 days. These patients will be followed up for improvement on the ground of clinical symptoms and serum bilirubin level and abdominal US for CBD stones.
  1. Improvement: If the stone spontaneously passes to the duodenum and CBD is clear completely from the stones proved by US, the patient will undergo laparoscopic cholecystectomy (LC) within 3 days.
  2. No improvement: the patient will undergo ERCP and then LC.
  Interventions: Procedure: conservative
- ERCP (endoscopic) (Active Comparator): 2- Patients in ERCP group will undergo ERCP and wide papillotomy and stone extraction directly then laparoscopic cholecystectomy (LC) within 3 days.cholecystectomy (LC) within 3 days.
  b- No improvement: the patient will undergo ERCP and then LC.
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: conservative — 1- Patients in conservative treatment group will receive medical treatment in the form of antibiotics (3rd generation cephalosporine), analgesics (NSAID eg Ibuprofen) and antispasmodics for 3 days. These patients will be followed up for improvement on the ground of clinical symptoms and serum bilirubin level and abdominal US for CBD stones.
  Other Names: G 1
  Arms: conservative
Procedure: ERCP — 2- Patients in ERCP group will undergo ERCP and wide papillotomy and stone extraction directly then laparoscopic cholecystectomy (LC) within 3 days.
  Other Names: G 2
  Arms: ERCP (endoscopic)

SUMMARY:
Evaluation of the best line of treatment of borderline CBD stones associated with gallbladder stones whether by conservative treatment or endoscopic stone extraction as regard complete clearance rate of the CBD stones followed by laparoscopic cholecystectomy. The secondary outcomes are overall complications related to each approach, technical difficulties and conversion rate during laparoscopic cholecystectomy and cost benefit relationship of each line of treatment.

DETAILED DESCRIPTION:
Enrolled patients in the study will be randomized to either conservative treatment or ERCP and stone extraction. The randomization process will be done using closed envelop method and will be withdrawn by a nurse in the outpatient clinic.

1. Patients in conservative treatment group will receive medical treatment in the form of antibiotics, analgesics and antispasmodics for 3 days. These patients will be followed up for improvement on the ground of clinical symptoms and serum bilirubin level and abdominal US for CBD stones.

   1. Improvement: If the stone spontaneously passes to the duodenum and CBD is clear completely from the stones proved by US, the patient will undergo laparoscopic cholecystectomy (LC) within 3 days.
   2. No improvement: the patient will undergo ERCP and then LC.
2. Patients in ERCP group will undergo ERCP and wide papillotomy and stone extraction directly then laparoscopic cholecystectomy (LC) within 3 days.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

1. CBD diameter less than 10mm.
2. Single or 2 stones in number.
3. Size of stone 5mm or less.
4. Serum bilirubin level less than 10 mg/dl .
5. SGPT, SGOT less than 300.
6. Associated gallbladder stones

Exclusion Criteria:

1. Previous cholecystectomy.
2. History of acute cholecystitis, pancreatitis, or cholangitis.
3. Previous history of endoscopic sphincterotomy.
4. Unfit patients for cholecystectomy.
5. No gallbladder stones.
6. Patients with altered GIT anatomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
complete clearance rate of the CBD stones | 30 DAYS
  complete clearance rate of the CBD stones

SECONDARY OUTCOMES:
overall complications | 30 DAYS
  pancreatitis
conversion rate during laparoscopic cholecystectomy | 1 day
  conversion rate during laparoscopic cholecystectomy

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El Nakeeb, MD, Principal Investigator — Mansoura University

REFERENCES:
- [Result] Hungness ES, Soper NJ. Management of common bile duct stones. J Gastrointest Surg. 2006 Apr;10(4):612-9. doi: 10.1016/j.gassur.2005.08.015. No abstract available. PMID 16627230
- [Result] Freitas ML, Bell RL, Duffy AJ. Choledocholithiasis: evolving standards for diagnosis and management. World J Gastroenterol. 2006 May 28;12(20):3162-7. doi: 10.3748/wjg.v12.i20.3162. PMID 16718834
- [Result] Samardzic J, Latic F, Kraljik D, Pitlovic V, Mrkovic H, Miskic D, Latic A, Delibegovic S. Treatment of common bile duct stones--is the role of ERCP changed in era of minimally invasive surgery? Med Arh. 2010;64(3):187-8. PMID 20645517
- See also: mansoura university — http://www.mans.edu.eg/